CLINICAL TRIAL: NCT01169064
Title: Topical Silver for Prevention of Wound Infection Post Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Topical Silver for Prevention of Wound Infection After Cesarean Delivery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed no statistical significance achieved.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kelly Bennett, Associate Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VUMFM-100785
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Wound Infection
Keywords: Wound infection prevention; Silver-containing surgical dressing; Cesarean delivery infection prevention
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silver-containing surgical dressing (Active Comparator): Self adhesive 4 x 10 dressing impregnated with nanocrystalline silver
  Interventions: Device: Silver-containing surgical dressing
- Cloth adhesive dressing (Active Comparator): Soft cloth adhesive wound dressing
  Interventions: Device: Cloth adhesive dressing

INTERVENTIONS:
Device: Silver-containing surgical dressing — Dressing placed over surgical incision and remain for 3-5 days
  Other Names: Acticoat
  Arms: Silver-containing surgical dressing
Device: Cloth adhesive dressing — Cloth adhesive dressing placed over surgical incision and remains for 3-5 days
  Other Names: Medipore
  Arms: Cloth adhesive dressing

SUMMARY:
A common concern in any surgical procedure is the occurrence of infection. Silver-containing treatments are popular and used in wound treatment; however, there is presently little evidence of the effectiveness of silver-containing treatment for the prevention of obstetrical wound infection. We plan to investigate the rate of infection in women experiencing cesarean sections at Vanderbilt University Medical Center (VUMC) by comparing the infection rate based on a randomized choice of silver-containing wound dressings to soft cloth adhesive wound dressings.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery with pfannenstiel incision

Exclusion Criteria:

* Incision other than pfannenstiel
* Silver allergy
* Inability to provide informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 475 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly A. Bennett, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Hospital, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 patients were removed from the study after consent but prior to study start, these participants did not meet inclusion / exclusion criteria
Period: Overall Study
Arm/Group | Silver-containing Surgical Dressing | Cloth Adhesive Dressing
Started | 239 | 236
Completed | 239 | 236
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age ranged from 16-45 but was not analyzed by treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Silver-containing Surgical Dressing | Cloth Adhesive Dressing | Total
Number analyzed (Participants) | 239 | 236 | 475
Age, Customized [Number; unit: years] — Age not recorded in several patients from both groups.
  years
    16-25 | 71 | 88 | 159
    26-35 | 143 | 113 | 256
    36-45 | 24 | 30 | 54
Sex/Gender, Customized [Number; unit: participants] — Women Only
  participants
    Women | 239 | 236 | 475
Race/Ethnicity, Customized [Number; unit: participants] — Race/Ethnicity was not captured on every patient.
  participants
    Caucasian | 155 | 156 | 311
    African American | 43 | 50 | 93
    Hispanic | 20 | 16 | 36
    Other | 17 | 10 | 27
Average BMI [Mean (Full Range); unit: kg/m^2] | 32.0 [28 to 36.3] | 32.8 [28.8 to 38.1] | 32.4 [28 to 38.1]
Tobacco use during pregnancy [Number; unit: participants]
  Yes | 49 | 41 | 90
  No | 190 | 195 | 385
No use of alcohol during pregnancy [Number; unit: participants] | 239 | 236 | 475

OUTCOME MEASURES:

1. Primary Outcome: Silver Treatment Efficacy
Description: As measured by number of patients with postop infections at 6 wks
Time Frame: 6 weeks postpartum
Measure: Number; unit: participants
Arm/Group | Silver-containing Surgical Dressing | Cloth Adhesive Dressing
Number analyzed (Participants) | 239 | 236
participants | 25 | 19
Statistical Analysis 1: Comparison: Silver-containing Surgical Dressing vs Cloth Adhesive Dressing; Test type: Superiority or Other; p = .365, Chi-squared

2. Secondary Outcome: Infection Rate Adjusted for Maternal BMI
Time Frame: 6 weeks postpartum
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Silver Dressing | Cloth Dressing
Number analyzed (Participants) | 239 | 236
percentage of participants | 10 [6.5 to 13.5] | 8 [4.1 to 11.9]
Statistical Analysis 1: Comparison: Silver Dressing vs Cloth Dressing; Test type: Superiority; p = .282, Mixed Models Analysis

3. Secondary Outcome: Patient Dressing Cost
Description: Total cost of dressings per group based on 1 dressing per patient
Time Frame: Postoperative
Measure: Number; unit: dollars
Arm/Group | Silver-containing Surgical Dressing | Cloth Adhesive Dressing
Number analyzed (Participants) | 239 | 236
dollars | 11,080.04 | 306.80

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Silver-containing Surgical Dressing: Self adhesive 4 x 10 dressing impregnated with nanocrystalline silver
  Silver-containing surgical dressing: Dressing placed over surgical incision and remain for 3-5 days
  No adverse events
- Cloth Adhesive Dressing: Soft cloth adhesive wound dressing
  Cloth adhesive dressing: Cloth adhesive dressing placed over surgical incision and remains for 3-5 days
  No adverse events
Arm/Group | Silver-containing Surgical Dressing | Cloth Adhesive Dressing
Serious Adverse Events (participants affected / at risk) | 3/239 | 3/236
Other Adverse Events (participants affected / at risk) | 25/239 | 19/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silver-containing Surgical Dressing (N=239) | Cloth Adhesive Dressing (N=236)
Readmission to hospital for Infection (Infections and infestations) | 3 (3) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silver-containing Surgical Dressing (N=239) | Cloth Adhesive Dressing (N=236)
Wound Infection (Infections and infestations) | 25 (25) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes